CLINICAL TRIAL: NCT00267956
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of CNTO 1275, a Fully Human Anti-IL-12 Monoclonal Antibody, Administered Subcutaneously, in Subjects With Active Psoriatic Arthritis
Brief Title: An Effectiveness and Safety Study of CNTO 1275 in Patients With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR006322; C0743T10 (Other: Centocor); 2005-003525-92 (EudraCT Number)
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis; CNTO 1275; Ustekinumab; Interleukin-23, IL-12, IL-23; Monoclonal antibodies
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CNTO1275 (ustekinumab) (Experimental): Group 1: Patients will receive CNTO 1275 63 mg at Weeks 0, 1, 2, and 3. At Weeks 12 and 16, patients will receive placebo to maintain the blind.
  Interventions: Drug: CNTO 1275 63 mg; Drug: Placebo
- Placebo (Placebo Comparator): Group 2: Patients will receive placebo at Weeks 0, 1, 2, and 3. At Weeks 12 and 16, patients will receive CNTO 1275 63 mg.
  Interventions: Drug: CNTO 1275 63 mg; Drug: Placebo

INTERVENTIONS:
Drug: CNTO 1275 63 mg — The patients will receive 90 mg (or 63 mg after filtration) subcutaneous injection on Weeks 0, 1, 2, and 3; Placebo subcutaneous injection on Weeks 12 and 16.
Drug: Placebo — The patients will receive placebo subcutaneous injection on Weeks 0, 1, 2, and 3; At weeks 12 and 16 the patients will receive CNTo1275 90 mg (or 63 mg after filtration) subcutaneous injection

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of CNTO 1275 (ustekinumab) in patients with psoriatic arthritis.

DETAILED DESCRIPTION:
This study is a randomized (the study drug is assigned by chance), double-blind (neither physician nor the patient knows the treatment that the patient receives), parallel-group (each group of patients will be treated at the same time), multicenter study to evaluate the effectiveness and safety of CNTO 1275 compared to placebo in the treatment of patients with active psoriatic arthritis. Patients will be randomized in 1:1 ratio to 1 of 2 treatment groups (CNTO 1275 63 mg and placebo). Patients will be randomly assigned to receive study medication up to Week 12 and will be followed through Week 36 to monitor safety and efficacy. Patients randomly assigned to placebo will crossover to receive CNTO 1275 63 mg at Weeks 12 and 16. Patients randomly assigned to CNTO 1275 will receive placebo at Weeks 12 and 16 to maintain the blind. The duration of participation for an individual patient in the study will be up to 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have had active psoriatic arthritis for at least 6 months prior to administration of first study injection
* Have an active plaque psoriasis (defined as a lesion of at least 2 cm in diameter), but not in armpits, on chest between breasts or groin
* Women of childbearing potential and all men must be using an effective method of birth control measures (eg, abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) and must agree to continue to use such measures until 12 months after receiving the last injection of study agent
* Have an active arthritis despite disease-modifying anti-rheumatic drugs (DMARD) such as leflunomide, gold, sulfasalazine, but not including methotrexate) or non-steroidal anti-inflammatory agents (NSAID) such as aspirin, ibuprofen, naproxen) therapy. DMARD therapy is defined as taking a DMARD for at least 3 months, or evidence of not tolerating DMARD. NSAID therapy is defined as taking an NSAID for at least 4 weeks
* If the patients are using methotrexate (MTX), they should have started treatment at least 3 months prior to the first administration of study agent and should have no serious toxic side effects attributable to MTX
* Have no signs or symptoms suggestive of active tuberculosis upon medical history, physical examination and chest X-ray

Exclusion Criteria:

* Have received DMARDs, other than methotrexate, within 4 weeks prior to the randomization visit
* Have used any biologic within the previous 3 months or 5 times the half-life of the biologic, whichever is longer
* Have received any oral, intravenous or intramuscular medications/treatments that could affect psoriasis (including, but not limited to, oral or injectable corticosteroids, retinoids, 1,25 dihydroxy vitamin D3 and analogues, psoralens, sulfasalazine, hydroxyurea, fumaric acid derivatives, or phototherapy) within 4 weeks of the randomization visit and/or have used topical medications/treatments that could affect psoriasis (eg, corticosteroids, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens) within 2 weeks of the randomization visit
* Have a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection (eg, bronchiectasis), recurrent urinary tract infection (recurrent pyelonephritis or chronic nonremitting cystitis), or open, draining, or infected skin wounds or ulcers
* Have a history of latent or active granulomatous infection, including tuberculosis (TB), histoplasmosis, or coccidioidomycosis, prior to screening
* Have current signs or symptoms of severe, progressive, or uncontrolled kidney, liver, blood, intestinal, hormonal, lung, heart, nervous, brain, or psychiatric disease
* Have any known cancer or have a history of cancer within the previous 5 years (with the following exception: have had basal cell carcinoma or squamous cell carcinoma in situ of the skin that has been treated, with no evidence of recurrence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2005-12; Primary Completion 2007-03 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (25):
- United States (12):
  - Macon, Georgia
  - Boise, Idaho
  - Normal, Illinois
  - Indianapolis, Indiana
  - Covington, Louisiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - New York, New York
  - Wilmington, North Carolina
  - Salt Lake City, Utah
- Canada (7):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Barrie, Ontario
  - Hamilton, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
- Denmark (3):
  - Aarhus C
  - Hellerup
  - København NV
- Finland (2):
  - Hus
  - Tampere
- Geneva, Switzerland

REFERENCES:
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Gottlieb A, Menter A, Mendelsohn A, Shen YK, Li S, Guzzo C, Fretzin S, Kunynetz R, Kavanaugh A. Ustekinumab, a human interleukin 12/23 monoclonal antibody, for psoriatic arthritis: randomised, double-blind, placebo-controlled, crossover trial. Lancet. 2009 Feb 21;373(9664):633-40. doi: 10.1016/S0140-6736(09)60140-9. Epub 2009 Feb 11. PMID 19217154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 146 participants were randomly assigned to receive either placebo or ustekinumab (CNTO 1275) at 24 sites in North America and Europe.
Groups:
- Placebo (CP): Controlled period (Week 0-12) - Placebo Group
- Ustekinumab x 4 (CP): Controlled period (Week 0-12) - Ustekinumab x 4 Group
- Placebo -> Ustekinumab (After CP): After Controlled period (Week 12-36) - receiving Placebo at Weeks 0, 1, 2, and 3 -> receiving ustekinumab at Week 12 and Week 16
- Ustekinumab x 4 (After CP): After Controlled period (Week 12-36) - receiving ustekinumab at Weeks 0, 1, 2, and 3 -> receiving Placebo at Week 12 and Week 16
Period: Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab x 4 (CP) | Placebo -> Ustekinumab (After CP) | Ustekinumab x 4 (After CP)
Started | 70 | 76 | 0 ("0" in column indicates this reporting group is not relevant to Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to Controlled Period.)
Completed | 57 | 72 | 0 | 0
Not Completed | 13 | 4 | 0 | 0
Not completed — Adverse Event | 4 | 1 | 0 | 0
Not completed — Lack of Efficacy | 4 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Withdrew consent | 3 | 1 | 0 | 0
Period: After Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab x 4 (CP) | Placebo -> Ustekinumab (After CP) | Ustekinumab x 4 (After CP)
Started | 0 ("0" in column indicates this reporting group is not relevant to after Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Controlled Period.) | 57 | 72
Completed | 0 | 0 | 52 | 70
Not Completed | 0 | 0 | 5 | 2
Not completed — Adverse Event | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrew consent | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group I: Placebo: Participants received subcutaneous (SC) placebo injection at Weeks 0, 1,2, and 3. At Week (Wk) 12 and Wk 16, placebo participants crossed over to receive ustekinumab (CNTO 1275) SC.
- Group II: Ustekinumab x 4: Participants received SC injection of ustekinumab 90 mg at Wk 0,1,2, and 3. At Wk 12 and Wk 16, participants received placebo SC to maintain the blind. After the first 36 participants were randomized, Centocor became aware that some vials of other study agents not used in this study contained black particulate matter and the filtration procedure was implemented. The resulting dose of ustekinumab after filtration was approximately 0.70 mL, equivalent to 63 mg.
- Total: Total of all reporting groups
Arm/Group | Group I: Placebo | Group II: Ustekinumab x 4 | Total
Number analyzed (Participants) | 70 | 76 | 146
Age Continuous [Mean (Standard Deviation); unit: years] | 47.1 (10.52) | 50.2 (11.23) | 48.7 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 37 | 45 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an American College of Rheumatology (ACR) 20 Response at Week 12
Description: ACR 20 response is an improvement of greater than or equal to 20 percentage in both tender and swollen joint count and in 3 to 5 assessments (patient's assessment of pain visual analog scale [VAS] with 0, no pain to 10, worst pain; patient's and physician's global assessment of disease activity VAS scales: overall disease activity [0, very well to 10, very poor and 0, no arthritis activity to 10, extremely active, respectively]; Health Assessment Questionnaire [HAQ]: 20-questions on life activities [0, no difficulty to 3, inability to perform a task]; C-reactive protein[CRP]).
Time Frame: Week 0 to Week 12
Population: Intent to treat. All participants randomized were included in the analysis according to the assigned treatment groups. Participant is considered a non- responder if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy or participant who have no data for all ACR components at Week 12.
Measure: Number; unit: Participants
Arm/Group | Group I: Placebo | Group II: Ustekinumab x 4
Number analyzed (Participants) | 70 | 76
Participants | 10 | 32
Statistical Analysis 1: Comparison: Group I: Placebo vs Group II: Ustekinumab x 4; Hypothesis: No difference between ustekinumab x 4 and placebo at a significant level of 0.05. Sample Size and power: With 70 partcipants in each treatment group, 5000 repetitions. Assuming a 20% ACR20 response in placebo participants regardless of prior anti-TNF exposure and a 35% ACR 20 and 45% ACR20 response in ustekinumab group for participants who had prior anti-TNF exposure, and who had no prior anti-TNF exposures, the power to detect the treatment difference is 0.85; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi-square — The study is designed to maintain a Type I error of 0.05 or less for the primary analysis; Stratified by subject's prior anti-Tumor Necrosis Factor (TNF) exposure status (Yes/No)

2. Secondary Outcome: Number of Participants With an American College of Rheumatology (ACR) 50 Response at Week 12
Description: ACR 50 response is an improvement of greater than or equal to 50 percentage in both tender and swollen joint count and in 3 to 5 assessments (patient's assessment of pain visual analog scale [VAS] with 0, no pain to 10, worst pain; patient's and physician's global assessment of disease activity VAS scales: overall disease activity [0, very well to 10, very poor and 0, no arthritis activity to 10, extremely active, respectively]; Health Assessment Questionnaire [HAQ]: 20-questions on life activities [0, no difficulty to 3, inability to perform a task]; C-reactive protein[CRP]).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group I: Placebo | Group II: Ustekinumab x 4
Number analyzed (Participants) | 70 | 76
Participants | 5 | 19
Statistical Analysis 1: Comparison: Group I: Placebo vs Group II: Ustekinumab x 4; Hypothesis: No difference between Group II and Group I at a significant level of 0.05; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel (CMH) chi-square — No multiplicity adjustment was made and nominal p-value was reported; Stratified by participant's prior anti-TNF exposure status (Yes/No)

3. Secondary Outcome: Number of Participants With an American College of Rheumatology (ACR) 70 Response at Week 12
Description: ACR 70 response is an improvement of greater than or equal to 70 percentage in both tender and swollen joint count and in 3 to 5 assessments (patient's assessment of pain visual analog scale [VAS] with 0, no pain to 10, worst pain; patient's and physician's global assessment of disease activity VAS scales: overall disease activity [0, very well to 10, very poor and 0, no arthritis activity to 10, extremely active, respectively]; Health Assessment Questionnaire [HAQ]: 20-questions on life activities [0, no difficulty to 3, inability to perform a task]; C-reactive protein[CRP]).
Time Frame: Week 12
Population: Intent to treat. All participant randomized were included in the analysis according to the assigned treatment groups. Participant is considered a non- responder if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy or participant who have no data for all ACR components at Week 12.
Measure: Number; unit: Participants
Arm/Group | Group I: Placebo | Group II: Ustekinumab x 4
Number analyzed (Participants) | 70 | 76
Participants | 0 | 8
Statistical Analysis 1: Comparison: Group I: Placebo vs Group II: Ustekinumab x 4; Hypothesis: No difference between ustekinumab x 4 and placebo at a significant level of 0.05; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel (CMH) chi-square — No multiplicity adjustment was made and nominal p-value was reported; Stratified by participant's prior anti-TNF exposure status (Yes/No)

4. Secondary Outcome: Change in Health Assessment Questionnaire (HAQ) at Week 12
Description: The HAQ is a 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area based on the worst score from the questions that pertain to that task. The HAQ score is determined by the average of the 8 scores.
Time Frame: Week 0 to Week 12
Population: Participants were included in the analysis according to the assigned treatment groups. Zero change is imputed if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy. Other missing data were not imputed.
Measure: Median (Inter-Quartile Range); unit: Scores on scale
Arm/Group | Group I: Placebo | Group II: Ustekinumab x 4
Number analyzed (Participants) | 64 | 75
Scores on scale | 0.00 [-0.25 to 0.13] | -0.25 [-0.50 to 0.00]
Statistical Analysis 1: Comparison: Group I: Placebo vs Group II: Ustekinumab x 4; Hypothesis: No difference between ustekinumab x 4 and placebo at a significant level of 0.05; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores — No multiplicity adjustment was made and nominal p-value was reported; Treatment and prior anti-TNF exposure (Yes/No) as factors in the model

5. Secondary Outcome: Number of Participants With Psoriasis Area and Severity Index (PASI) Score of 75 Percent at Week 12
Description: Number of participants achieving greater than or equal to 75 perccentage mprovement PASI at Week 12. PASI is widely used tool for the measurement of severity of psoriasis. This is a test of how bad person's psoriasis is. The combine redness, scaling, and thickness, as well as overall body involvement determine the PASI score. The scale ranges from 0 (best) to 72 (worst).
Time Frame: Week 12
Population: All participants randomized with baseline ≥ 3% body surface area (BSA) psoriatic involvement and with evaluable measurement are included in the analysis according to the assigned treatment groups. Participant is considered a non- responder if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy.
Measure: Number; unit: Participants
Arm/Group | Group I: Placebo | Group II: Ustekinumab x 4
Number analyzed (Participants) | 55 | 63
Participants | 3 | 33
Statistical Analysis 1: Comparison: Group I: Placebo vs Group II: Ustekinumab x 4; Hypothesis: No difference between ustekinumab x 4 and placebo at a significant level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi-square — No multiplicity adjustment was made and nominal p-value was reported; Stratified by participant's prior anti-TNF exposure status (Yes/No)

6. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) at Week 12
Description: Change in Dermatology Life Quality Index (DLQI) from baseline at Week 12. The DLQI is a 10 item questionnaire, is designed to assess the impact of the disease on a participant's quality of life, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The score ranges from 0 (better quality of life) to 30 (worse quality of life).
Time Frame: Week 0 to Week 12
Population: All participants randomized with baseline ≥ 3% body surface area psoriatic involvement were included in the analysis according to the assigned treatment groups. Zero change is imputed if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy. Other missing data were not imputed.
Measure: Median (Inter-Quartile Range); unit: Scores on scale
Arm/Group | Group I: Placebo | Group II: Ustekinumab x 4
Number analyzed (Participants) | 55 | 63
Scores on scale | 0.00 [-4.0 to 2.0] | -6.0 [-14.0 to -3.0]
Statistical Analysis 1: Comparison: Group I: Placebo vs Group II: Ustekinumab x 4; Hypothesis: No difference between ustekinumab x 4 and placebo at asignificant level of 0.05; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores — No multiplicity adjustment was made and nominal p-value was reported; Treatment and prior anti-TNF exposure (Yes/No) as factors in the model

ADVERSE EVENTS:
Time Frame: 36 weeks
Description: 2 participants discontinued study agent during the controlled period (CP) but had follow-up after CP and hence are included in the tables of frequent adverse events and serious adverse events after CP.
Groups:
- Ustekinumab x 4 (CP): Controlled period (Week 0-12) - Ustekinumab (CNTO 1275) x 4 Group
Arm/Group | Placebo (CP) | Ustekinumab x 4 (CP) | Placebo -> Ustekinumab (After CP) | Ustekinumab x 4 (After CP)
Serious Adverse Events (participants affected / at risk) | 3/70 | 0/76 | 4/57 | 2/74
Other Adverse Events (participants affected / at risk) | 19/70 | 29/76 | 19/57 | 24/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=70) | Ustekinumab x 4 (CP) (N=76) | Placebo -> Ustekinumab (After CP) (N=57) | Ustekinumab x 4 (After CP) (N=74)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=70) | Ustekinumab x 4 (CP) (N=76) | Placebo -> Ustekinumab (After CP) (N=57) | Ustekinumab x 4 (After CP) (N=74)
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 2 | 3 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 2
Influenza (Infections and infestations) | 4 | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 2 | 8 | 4 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 10 | 6 | 7
C-reactive protein increased (Investigations) | 1 | 1 | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4
Headache (Nervous system disorders) | 4 | 5 | 2 | 1

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse event (NAE) excludes patients who only had NAE that occured in <= 5% of patients. This information may vary from existing approved labeling and publications due to the requirements of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.